CLINICAL TRIAL: NCT06177834
Title: Comparison of Alisklamp and Dorsal Slit Sleeve Circumcision: A Randomized Controlled Trial
Brief Title: Alisklamp and Dorsal Slit Sleeve Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Azizoğlu (Other)
Responsible Party: Sponsor-Investigator, Mustafa Azizoğlu, MD, Necmi Kadıoğlu Hospital
Organization: Necmi Kadıoğlu Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NecmiKadiogluH
Record Dates: First submitted 2023-11-24; First posted 2023-12-20 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Circumcision

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical dorsal slit circumcision technique (Active Comparator): In this group, the patients who will operated with dorsal sleeve slit circumcision technique.
  Interventions: Other: Dorsal slit circumcision technique
- Alisklamp (Experimental): In this group, the patients who will operated with Alisklamp technique.
  Interventions: Device: Alisklamp

INTERVENTIONS:
Device: Alisklamp — Alisklamp
  Arms: Alisklamp
Other: Dorsal slit circumcision technique — In this group, included the patients who will operated with dorsal slit circumcision technique
  Arms: Classical dorsal slit circumcision technique

SUMMARY:
In this study the plan is to compare the circumcision performed with Alisklamp versus Dorsal Slit Sleeve method in terms of age, co-existing health conditions, surgery time, recovery period, tissue edema and bleeding, postoperative infection, wound healing, wound dehiscence, skin tunnel, and overall complications.

DETAILED DESCRIPTION:
The study compares two circumcision techniques in children: the dorsal sleeve slit method and the alisclamp method. The dorsal sleeve slit technique, conducted under local anesthesia for about 20-30 minutes, involves cutting the penile skin dorsally, removing excess skin and prepuce, and suturing with 5/0 vicryl. The alisclamp method, also under local anesthesia, entails retracting the penile skin, placing a clamp, excising excess prepuce, and sending the patient home. The clamp is removed after 48 hours without anesthesia, with the total procedure lasting under 5 minutes. This research assesses these methods based on factors like age, co-existing health conditions, surgery time, recovery period, tissue edema and bleeding, postoperative infection, wound healing, wound dehiscence, skin tunnel, and overall complications.

ELIGIBILITY:
Inclusion Criteria:

male patients between 0-2 years and 6-18 years

Exclusion Criteria:

2-6 years, several penil chordee, hypospadias, previous penil surgery

Ages: 1 Minute to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male
Enrollment: 180 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Healing time | 2 weeks
  Healing time
infections | 2 weeks
  wound infections
wound dehiscence | 2 weeks
  wound dehiscence
skin tunnel | 1 month
  presense of the number of skin tunnel

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Azizoğlu, Principal Investigator — Necmi Kadıoğlu State Hospital
Locations (1):
- Mustafa Azizoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No